CLINICAL TRIAL: NCT02665767
Title: A Feasibility Study of Telementoring for Identifying the Appendix Using Smartphone-based Telesonography
Brief Title: Telementoring for Identifying the Appendix Using Telesonography
Acronym: TIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Fellowship, Emergency Medincine, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hanyang University
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Appendix, Ultrasonography
Keywords: Telesonography, Appendix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On-site sonography (No Intervention): The subjects(n=15) performed ultrasonography for the identification of the appendix under mentoring by an onsite expert.
- Smartphone-based Telesonography (Active Comparator): The subjects(n=15) performed ultrasonography for the identification of the appendix under mentoring by an offsite expert.
  Interventions: Device: Smartphone-based Telesonography

INTERVENTIONS:
Device: Smartphone-based Telesonography — The 30 participating examiners were randomly divided into two groups. In phase one, group A performed ultrasonography under onsite mentoring and group B performed the same procedure under remote mentoring. Each examiner was randomly assigned one expert and three SPs for phase one. Four weeks later, they were partnered with the same expert and SPs to whom they had been assigned in phase one and performed the procedure under the other type of mentoring (phase two). The examination order of the SPs was randomly assigned by choosing a number between one and six (1: A-B-C, 2: A-C-B, 3: B-A-C, 4: B-C-A, 5: C-A-B, 6: C-B-A) in each phase.
  Arms: Smartphone-based Telesonography

SUMMARY:
The investigators investigated the feasibility of the clinical application of novice-practitioner-performed/offsite-mentor-guided ultrasonography for identifying the appendix.

DETAILED DESCRIPTION:
A randomized cross-over study was conducted using a telesonography system that can transmit the ultrasound images displayed on the ultrasound monitor(ultrasound sequence video) and images showing the practitioner's operations(background video) to a smartphone without any interruption in motion over a Long Term Evolution (LTE) network. Thirty novice practitioners were randomly assigned to two groups. The subjects in group A (n=15) performed ultrasonography for the identification of the appendix under mentoring by an onsite expert, whereas those in group B (n=15) performed the same procedure under mentoring by an offsite expert.

Each subject performed the procedure on three simulated patients. After a four-week interval, they performed the procedure again under the other type of mentoring. A total of 90 ultrasound examinations were performed in each scenario. The primary outcomes were the success rate for identifying the appendix and the time required to identify the appendix.

ELIGIBILITY:
Inclusion Criteria:

* Without any experience in ultrasonography

Exclusion Criteria:

* Subjects who do not want to participate
* Subjects who has eye pain or any eye problem
* Subjects who has wrist pain

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Success rate | 8 months
  "Success" is meaning of identifying appendix in 10 minutes.

SECONDARY OUTCOMES:
Time to identifying appendix | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: YOONJE LEE, M.D., Principal Investigator — Departement of Emergency Medicine, Hanyang University Guri Hospital
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea